CLINICAL TRIAL: NCT06643754
Title: A Phase I/II Clinical Study on the Safety, Tolerability, Pharmacokinetics, and Efficacy of SHR-3276 Injection in Patients With Advanced Malignant Tumors
Brief Title: A Clinical Study of SHR-3276 for Injection in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-3276-101
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Single arm study of SHR-3276
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-3276 for Injection will be administrated per dose level in which the patients are assigned. (Experimental)
  Interventions: Drug: SHR-3276

INTERVENTIONS:
Drug: SHR-3276 — Dose Escalation: SHR-3276 will be administered intravenously. 4 dose levels are preset.
  Dose Expansion: 2 to 3 dose cohorts will be selected for dose expansion stage.
  Indication Expansion: Indications will be selected to evaluate preliminary efficacy.

SUMMARY:
This study is an open-label, multicenter Phase I/II clinical trial to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-3276 for injection in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to sign a written informed consent；
2. Age 18-70 years old (including both ends), both male and female；
3. Pathologically confirmed advanced malignant tumors that have failed sufficient standard treatment or have no effective standard treatment plan；
4. Existence of measurable lesions；
5. ECOG score: 0-1；
6. Expected survival time ≥ 12 weeks；
7. The functional level of the major organs must meet the requirements；
8. Fertile female patients must have a serum pregnancy test within 7 days before the first medication and the result is negative; And must be non-lactating.

Exclusion Criteria:

1. Central nervous system metastasis or meningeal metastasis with clinical symptoms;
2. Spinal cord compression that has not been treated radically by surgery and/or radiotherapy；
3. Patients with uncontrolled tumor-related pain as judged by the investigator
4. A third space effusion with uncontrolled pleural effusion, pericardial effusion, or peritoneal effusion, as determined by the investigator；
5. Systemic antitumor therapy was administered within 28 days prior to treatment in the first study；
6. Surgical procedures requiring tracheal intubation and general anesthesia were performed within 28 days prior to the initial study, or elective surgery was expected during the trial period；
7. Serious drug-related adverse reactions during previous immune checkpoint inhibitor therapy；
8. Has unresolved toxicities from previous anticancer therapy, defined as toxicities not yet resolved to NCI-CTCAE version 5.0 grade ≤ 1；
9. Live attenuated vaccines were used within 28 days prior to administration in the first study or were expected to be required during the study treatment；
10. Systemic immunosuppressive therapy was administered within 14 days prior to the first study
11. Arterial/venous thrombosis events occurred within 3 months prior to initial administration
12. Patients with clinical significant lung disease;
13. Patients with history of autoimmune diseases;
14. The first study studied any other malignancy within 5 years prior to medication
15. A known history of severe allergic reactions to the investigational drug and its principal formulation ingredients；
16. Have a history of immune deficiency or organ transplantation；
17. Other serious accompanying illnesses, which, in the investigator's assessment, could seriously adversely affect the safety of the treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | up to 3 years
MTD | up to 6 months
RP2D | up to 1 year

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | up to 3 years
Maximum concentration (Cmax) | up to 3 years
Receptor Occupancy（OR） of SHR-3276 | up to 3 years
Anti-drug antibody (ADA) of SHR-3276 | up to 3 years
Objective response rate (ORR) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years
Duration of response (DoR) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years
Disease control rate (DCR) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years
Progression free survival（PFS） | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years
Overall survival (OS) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of PLA Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided